CLINICAL TRIAL: NCT06785961
Title: Healing Assessment of External Inflammatory Root Resorption After Revascularization Technique of Avulsed Permanent Central Incisor (Case Study)
Acronym: (EIRR)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Abdelrhaman Reda Elshair, Teaching assistant at badr university in cairo, Badr University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUC-IACUC-241020-113
Record Dates: First submitted 2024-12-08; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Avulsion
MeSH Terms: conditions — Fractures, Avulsion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single- arm (Experimental): Case study
  Interventions: Procedure: Regeneration of traumatic tooth

INTERVENTIONS:
Procedure: Regeneration of traumatic tooth — Revascularization is a new treatment method for immature necrotic , pulp revascularization allows also the stimulation of the apical development and the root maturation of immature teeth ( growth and thickening of dentinal walls ).

SUMMARY:
Evaluate the healing of external root resorption of replanted avulsed permanent maxillary central incisor after revascularization.

DETAILED DESCRIPTION:
Healing assessment of external inflammatory Root Resorption after Revascularization Technique of Avulsed permanent Central Incisor (Case study)

ELIGIBILITY:
Inclusion Criteria:

* traumatic teeth
* external inflammatory root resorption

Exclusion Criteria:

-

Min Age: 11 Months | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Measure amount of bone healing and root formation by using cone beam computed tomography (CBCT) | 18 months
  Measure amount of bone healing and root formation by using measuring tool cone beam computed tomography (CBCT) By using measuring unit hounsfield unit (HU)

SECONDARY OUTCOMES:
Measuring pain by using the numeric pain rating scale | 18 months
  Measuring pain by using the numeric pain rating scale, through patient is asked to make three pain rating, the average of three ratings was used to represent the patient's level of pain (0 none) (1-3 mild) (4-6 moderate) (7-10 severe)
Pulp test to assess the vitality or health of the dental pulp | Every 6 months
  Pulp test to assess the vitality or health of the dental pulp through measuring tool thermal pulp test :applied to the tooth to assess the response. The unit of measurement here is typically °C (degrees Celsius) .

CONTACTS AND LOCATIONS:
Locations (1):
- Badr university in Cairo, Badr, Cairo Governorate, Egypt